CLINICAL TRIAL: NCT02817958
Title: Prospective Phase II Study Evaluating a Multimodal Care of Inguinal Node Metastasis in Squamous Cell Carcinoma of the Penis by Bilateral Lymphadenectomy and Chemotherapy TIP
Brief Title: Evaluation of Lymphadenectomy and Chemotherapy TIP on Inguinal Lymph Nodes in Squamous Cell Carcinoma of the Penis
Acronym: MEGACEP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0160/1406; AFU-GETUG 25 (Other: Unicancer); 2014-004678-41 (EudraCT Number)
Record Dates: First submitted 2016-05-24; First posted 2016-06-29 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Penile Cancer; Squamous Carcinoma
Keywords: inguinal lymph nodes; penile cancer; squamous; TIP chemotherapy
MeSH Terms: conditions — Penile Neoplasms; Carcinoma, Squamous Cell | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-Adjuvant Chemotherapy TIP (Experimental): Lymphadenectomy (+/- sentinel node) + adjuvant chemotherapy TIP modified bilateral lymphadenectomy 4 cycles every 21 days
  Interventions: Drug: Chemotherapy TIP
- B-Neoadjuvant Chemotherapy TIP (Experimental): fine needle biopsy or sentinel node + neoadjuvant chemotherapy TIP followed by a lymphadenectomy modified bilateral lymphadenectomy 4 cycles every 21 days
  Interventions: Drug: Chemotherapy TIP

INTERVENTIONS:
Drug: Chemotherapy TIP — Paclitaxel, ifosfamide, and cisplatin
  Other Names: Chemotherapy TIP (paclitaxel, ifosfamide et cisplatine)

SUMMARY:
Squamous cell carcinoma of the penis is a rare tumor in Europe, whose prognosis and survival are influenced by metastatic lymph node involvement. Its frequency in France is estimated at less than 1% of human cancers. This spread follows a sequential process via the superficial and deep inguinal lymph nodes and then to the pelvic lymph nodes before metastatic dissemination.

The management of inguinal areas is the cornerstone of penile cancer. It is curative in about 80% of patients with 1 or 2 inguinal metastases. 5-years overall survival was on average 85% for pN0 patients and 40% for pN+ patients. For pN+ patients, 5-year overall survival was 70 to 80% for pN1 (only 1 lymph node invasion), 30 to 40% for pN2, and 0 to 10% for pN3.

The risk of local recurrence is 5-10% for pN0 and 20-30% for pN+ after local treatment by lymphadenectomy alone without chemotherapy. The average time to recurrence was 10 months. Disease-free survival at 5 years is 75-85% for pN0 and 30-45% for pN+. Its indication depends on clinical examination (presence or absence of lymph nodes palpated) and the risk of nodal disease (≥pT1bG2).

Currently, a fine needle biopsy is the best clinical diagnosis method because it is a simple, low risk, and possible in consultation. When the result is positive, it allows an early dissection. Single or double fine needle biopsy will be used in cN+ patients. For patients at risk of lymp nodes involvement (cN0 and ≥pT1B or G2), the sentinel node diagnosis may be followed by modified or bilateral lymphadenectomy.

Although lymphadenectomy alone has a curator action, it sometimes remains insufficient in patients with metastatic lymph node involvement. Therefore it seems important to develop a multimodal approach in the management of these patients in order to increase the response rate to treatment and survival.

From a Phase II trial conducted on 30 patients, the combination TIP (paclitaxel, ifosfamide, and cisplatin) appears to have an efficacy / toxicity acceptable.

The TIP protocol has therefore been chosen for this trial as adjuvant or neo-adjuvant treatment in patients with high risk of lymph nodes involvement (cN0 and ≥pT1B or G2), and with inguinal mobile palpated lymph nodes (cN+) respectively, after lymph nodes involvement proven (pN+).

ELIGIBILITY:
Inclusion Criteria:

1. penile tumor histologically proven whatever the initial treatment of penile tumor: amputation or conservative surgery or brachytherapy,
2. Mobile palpated lymph nodes (stage cN1 and cN2) whatever the T stage, Or If no palpated lymph nodes (cN0), patients with nodes involvement risk ≥pT1b and / or Grade 2,
3. Metastatic lymph node involvement,
4. Patients M0 or Mx,
5. Age ≥18 ans,
6. Eastern Cooperative Oncology Group (ECOG) 0-1,
7. Leucocytes ≥1.5 g/L,
8. Hemoglobin ≥9 g/dL,
9. Platelets ≥100 000/mm³,
10. Normal calcemia and kaliemia,
11. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤1.5 upper limit of normal (ULN) ; total bilirubin ≤1.5 ULN (3 ULN in case of Gilbert disease); alkaline phosphatase (ALP) <2 ULN,
12. Creatinine clearance ≥60 mL/min (MDRD method),
13. Left ventricular ejection fraction (LVEF) >50%,
14. Patients having received, read the information note and signed consent,
15. Reproductive age patients agreeing to use two methods of birth control (one for the patient and one for the partner) for the duration of the study and for 6 months after the last dose of treatment,
16. Patients able to comply with the protocol requirements (scheduled visits, treatment plan, clinical, paraclinical, biological and other procedures of the Protocol),
17. Patients undergoing a social security scheme.

Exclusion Criteria:

1. Fixed inguinal lymph nodes (cN3),
2. Iliac lymph nodes (cN3),
3. Patients pN3,
4. prior chemotherapy for squamous cell carcinoma of the penis,
5. Against-indication for chemotherapy or known hypersensitivity to cisplatin, ifosfamide or paclitaxel,
6. Patients treated with phenytoin,
7. Patients with hearing loss >Grade 1 (CTCAE V4.03),
8. Patients with cardiopulmonary disease-indicating against overhydration,
9. History of cancer within 5 years prior to inclusion in the trial other than cutaneous basal cell,
10. Patient received a live attenuated vaccine within 30 days prior to inclusion,
11. Patients already included in another clinical trial or receiving an experimental treatment within 30 days prior to inclusion in the trial,
12. Patients deprived of their liberty or under court protection including guardianship,
13. Severe systemic disease or uncontrolled or any other chronic or acute illness that is incompatible with the patient's participation in the trial according to investigator,
14. immunocompromised patients including with known seropositivity (HIV),
15. Patients with mental impairment which prevents the understanding of the protocol or having a psychological state, family, sociological or geographical conditions that would not allow compliance with the protocol and the planned follow-up or any condition which, according to the investigator, would prevent participation patient tested. These conditions should be assessed before inclusion of patients.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2016-10-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
survival without locoregional lymph node recurrence | 24 months
  checked by inguinal ultrasound

SECONDARY OUTCOMES:
Complete response rate for patients in neoadjuvant chemotherapy | 6 months
  lack of residual tumor post surgical histopathology
Survival without locoregional lymph node recurrence | 3 years
  time between inclusion and locoregional recurrence or last evaluation
Survival without metastasis | 3 years
  time between inclusion and the date of occurrence of metastases
Specific survival | 3 years
  time between inclusion and date of death from penile cancer or treatment-related complication
Overall survival | 3 years
  time between inclusion and the death regardless of cause
Acute and late toxicity during the study | Throughout study completion, up to 3 years
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 4.03 (NCI-CTCAE v4.03) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3
  = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
Quality of life questionnaire - Core 30 (QLQ-C30) | baseline, during treatment (C3J42), 6 month, 1 year
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials. The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Rigaud, Professor, Principal Investigator — Nantes University Hospital
Locations (17):
- France (17):
  - ICO-Paul Papin, Angers
  - Chr Besancon, Besançon
  - Hôpital SAINT ANDRE, Bordeaux
  - Centre FRANCOIS BACLESSE, Caen
  - Chru Gabriel Montpied, Clermont-Ferrand
  - Ch de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Chu Lyon Sud, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut de Cancerologie de Lorraine, Nancy
  - Clinique Urologique- Chu Hotel Dieu, Nantes
  - Institut de Cancerologie Du Gard - Centre Oncogard, Nîmes
  - Hopital Saint Louis, Paris
  - Chu de Rouen, Rouen
  - ICO-René Gauducheau, Saint-Herblain
  - Hopitaux Universitaires de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.